CLINICAL TRIAL: NCT04674839
Title: The Impact of MS-20 on Gut Microbiota Composition, Sera Endotoxin, Trimethylamine N-oxide, Metabolism and Immune Cell Profiling in Adult Individuals
Brief Title: The Impact of MS-20 on Gut Microbiota Composition in Adult Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS20CLIIS01
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Microbiota

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS-20 (Experimental): 8 ml/day for 8 weeks
  Interventions: Drug: MS-20
- Placebo (Other): 8 ml/day for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MS-20 — fermented soymilk product
  Arms: MS-20
Other: Placebo — No active ingredient
  Arms: Placebo

SUMMARY:
MicrSoy-20 (MS-20), a fermented soymilk product, has been approved as an Over the counter (OTC) drug in 2011. The therapeutic effect of MS-20 is to ameliorate symptoms such as fatigue and loss of appetite caused by cancer chemotherapy. Animal study revealed orally administration of MS-20 daily for 4 weeks altered the gut microbiota composition in mice. In addition, MS-20 could activate dendritic cell and improve immunotherapy response rate. Thus, it was hypothesis that MS-20 improves host immune activity thus ameliorate fatigue and increase weight is through alteration the gut microbiota composition.

In this study, the ability of MS-20 in modulating gut microbiota and the subset of microbiome to be altered by MS-20 was investigated.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, investigator-initiated randomized trial to evaluate the impact of MS-20 on gut microbiota composition and abundance in healthy people. Approximately 100 subjects who meet the criteria of this study are planned to be enrolled. Eligible subjects will be randomized to receive placebo or MS-20 in a 1:1 ratio with 50 subjects in each arm.

The study comprises of a 7 days screening period, a 8-week treatment period and a 8-week follow-up period. Eligible subjects will receive MS-20 or placebo every day during the treatment period. Participants should not use any probiotics and prebiotics during the trial. In addition, All medications (especially antibiotics) should be recorded and documented, however, fluoroquinolones and vancomycin will be banned during the trial.

The fecal gut microbiota, serum, and urea were collect at indicated time. The gut microbiota composition, gut microbiota metabolite, and serum biochemical items will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 20 and 65 years old.
2. The subject is able to provide written informed consent by himself/herself and agrees to comply with all protocol requirements.
3. The subject agrees to comply with the following two requirements:

   1. comply with all follow-up visit requirements according to the trial protocol.
   2. comply with all requirement regarding fecal samples collection, storage and delivery according to the trial protocol.

Exclusion Criteria:

1. The subject has soybean allergy.
2. The subject is pregnant or lactating.
3. The subject has received or is receiving chemotherapy.
4. The subject has received any antibiotic, antifungals or antivirals (excluding topical agents and antiviral prophylaxis for hepatitis B virus) within 30 days prior to visit 1 .
5. The subject has a clinically significant, currently active or underlying diarrhea (soft or loose stools more than three times in 24 hours) of infectious etiologies.
6. The subject has received any steroids, immunosuppressant or anti-inflammation drugs within 30 days prior to visit 1.
7. The subject has received probiotics or prebiotics 30 days prior to visit 1
8. The subject who has been diagnosed a chronic kidney disease, chronic gut inflammatory disease, cancer, or autoimmune disease within 1 year before participating this study.
9. Alcohol abuse, and smoking abuse.
10. The subject has active inflammatory bowel disease or gastric ulcer.
11. The subject currently is participating in studies involving other investigational drugs, medical devices, functional foods, or cosmetic.
12. The subject is considered by the investigator as not suitable for the trial.
13. The subject is judged by the investigator as not suitable for the trial due to concerns about possible non-compliance or severe concomitant illnesses.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Gut microbiota from baseline to 8th week | baseline to 8th week
  The composition, abundance and diversity of gut microbiota change from baseline in subjects treated with MS-20 or Placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Microbio Group, Taipei, Taiwan